CLINICAL TRIAL: NCT03264911
Title: Group A Streptococcal Pharyngitis: Six Days Amoxicillin, oR Six Days Placebo in Children Between 3 and 15 Years Old:a Randomized, Double Blinded, Multicentred, Non-inferiority Trial
Brief Title: Group A Pharyngitis in Children: The GASPARD Study
Acronym: GASPARD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klara Posfay-Barbe (Other)
Collaborators: Gertrude Von Meissner Foundation (Other); Recherche et Développement des HUG (Unknown); Société académique de Genève (Unknown)
Responsible Party: Sponsor-Investigator, Klara Posfay-Barbe, Head of Pediatric Infectious Diseases, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GASPARD
Record Dates: First submitted 2017-08-15; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Group A Streptococcal Pharyngitis
Keywords: pharyngitis; amoxicillin
MeSH Terms: conditions — Pharyngitis | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: prospective, randomized, interventional, placebo-controlled, double-blinded, multicentric clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- amoxicillin (Active Comparator): Children will be randomized to receive, after consent to the study, an antibiotic (amoxicillin approximately 50 mg/kg/day) orally, twice a day for 6 days.
  Interventions: Drug: Amoxicillin or Placebo
- Placebo arm (Placebo Comparator): Children will be randomized to receive, after consent to the study, a placebo orally, twice a day for 6 days.
  Interventions: Drug: Amoxicillin or Placebo

INTERVENTIONS:
Drug: Amoxicillin or Placebo — Children will be randomized to either 6 days of amoxicilline or 6 days of placebo treatment

SUMMARY:
Evaluate the necessity to treat with antibiotics GAS pharyngitis in children in Switzerland. The null hypothesis is that antibiotic treatment is not necessary for GAS pharyngitis in this population.

DETAILED DESCRIPTION:
All children between 3 -15 years old with clinical symptoms suggestive of pharyngitis (Mc Isaac score ≥3) and a microbiological test (rapid antigen detection) positive for group A Streptococcus (GAS) will be included in the study. In order to assess the strain of GAS as well as to identify co-infected children with respiratory virus, a throat culture and a nasopharyngeal swab will be performed, as well as a standard questionnaire and a standard physical exam. At this time, children will be randomized to either 6 days of amoxicilline or 6 days of placebo treatment. During the treatment period, the investigators will ask the parents/legal guardians of the patients to pay close attention to the evolution of the symptoms (fever, pain, exudates…) as well as the treatment's adverse event, and to report their presence or absence in a dairy form. At day three after initiation of treatment, a standardized clinical evaluation will be completed by phone to identify if the patient still has symptoms of pharyngitis or signs of suppurative complications. One month after the inclusion in the study, a throat culture, a standardized questionnaire as well as a clinical evaluation will be performed to identify if the patient has or had signs of non-suppurative complications and non-resolving infection. Six month and one year after inclusion, a phone call will evaluate the possible relapses, recurrences and complications of GAS infection with a standardized questionnaire. GAS strains will be analyzed to identify their unique fingerprint and viral coinfections will be reported to possibly identify cofactors for increased complication rates.

ELIGIBILITY:
Inclusion Criteria:

* 3 -15 years old
* Clinical symptoms suggestive of pharyngitis with MC Isaac score ≥3
* Rapid-antigen detection test (RADT) positive for GAS-
* Signed informed parental/patient consent form

Exclusion Criteria:

* Hypersensitivity to B-lactams
* concomitant disease which must be treated with antibiotics
* chronic disease-Immunocompromised
* Antibiotics within 72 h
* history of ARF,scarlet fever,impetigo,acute glomerulonephritis
* Family history of ARF
* Complicated pharyngitis

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Non inferiority | up to 1 month
  Duration of fever and other clinical signs/symptoms in not treated children versus treated

SECONDARY OUTCOMES:
Number of consultations for pharyngitis | 1 year
  To evaluate number of repeated consultations with pediatrician due to non-resolving/recurrent symptoms
suppurative complications | 1 year
  to evaluate rates of suppurative complications (acute otitis media-sinusitis-quinsy-cellulitis-impetigo) of GAS infections
non-suppurative complications | 1 year
  to evaluate rates of non-suppurative complications(ARF-glomerulonephritis-scarlet fever) of GAS infections
eradication | 1 month
  to evaluate bacteriological eradication rates of the initial pathogen
co-infections | at inclusion
  to discover if respiratory viruses are detected as co-infections in children with GAS pharyngitis upon initial presentation and during a recurrent episode
GAS strains | 1 month
  to investigate the biology and genetic structure of GAS strains in Switzerland.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Posfay-Barbe, Principal Investigator — Coordinator
Locations (1):
- Children's Hospital of Geneva (HUG), Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gualtieri R, Verolet C, Mardegan C, Papis S, Loevy N, Asner S, Rohr M, Llor J, Heininger U, Lacroix L, Pittet LF, Posfay-Barbe KM. Amoxicillin vs. placebo to reduce symptoms in children with group A streptococcal pharyngitis: a randomized, multicenter, double-blind, non-inferiority trial. Eur J Pediatr. 2024 Nov;183(11):4773-4782. doi: 10.1007/s00431-024-05705-1. Epub 2024 Aug 31. PMID 39215861